# Informed Consent Form

Study Title: Social Media Indoor Tanning Study

NCT03834974

# Information Sheet for Participation in a Research Study



Principal Investigator: Sherry Pagoto, Ph.D. Study Title: Social Media and Young Adults Sponsor: The National Institutes of Health

### Overview of the Research:

You are being asked to provide consent to participate in a research study. Participation is voluntary. You can say yes or no. If you say yes now you can still change your mind later. Some key points to consider are summarized in this overview, but you should consider all of the information in this document carefully before making your decision.

- This research is being done to deliver health information on Twitter and Facebook, specifically about lifestyle and mental wellbeing. We are doing a 4-week contest, which includes participants making the posts about the health information with weekly chances to win a gift card as well as compensation for creating each post. We will give you the health information to put into your posts.
- Participation includes an initial survey to see if you are eligible, a brief conversation to tell you about the study, a short survey to gather information about your lifestyle and wellbeing, a 30-minute webinar to talk about research and participation, 4 weeks of a social media contest, and a final survey to gather your opinions on your participation.
- Participation will involve approximately 2 and a half hours of your time over the next 6 weeks.
- Compensation is in the form of Amazon gift cards and includes \$10 for each post (up to \$60), a chance to win \$50 in each of the 4 week of the contest, and \$50 at the end of the study. You can also receive \$25 if you refer a friend who enrolls in the study.
- A possible risk of participating is release of confidential information. Some of the questions on the surveys may also cause you to feel upset. You may choose to not answer any question you do not wish to answer. Risks are described in more detail later in this form.
- There may also be benefits of participation such as increased awareness of physical and mental wellbeing.

### Introduction

You are being asked to participate because you are a regular social media user interested in topics related to health, lifestyle, and physical and mental wellbeing.

# Why is this study being done?

The purpose of this research is to test the best way to provide accurate information on physical and mental wellbeing using Twitter and Facebook.

## What are the study procedures? What will I be asked to do?

This is an online-only study. If you would like to take part in this research, your participation will last approximately 6 weeks and will include:

- A screening phase
- 4-week contest in which you create posts on certain topics which will appear in our Center's Twitter and Facebook feed
- Online survey before the study and after the contest

### Screening phase:

The screening phase includes an initial 5-minute online survey, a 10-minute telephone conversation with our study staff, a second online survey lasting about 15 minutes. Once we have determined that you are eligible, you will be randomized into the study to determine which feed your posts will go on.

#### Webinar:

After randomization, you will attend at 30-minute webinar so we can explain the study procedures in more detail, give you some background information on the social media feed your posts will go on, and to explain how the contest will work.

#### Contest:

The contest last for 4 weeks and includes creating 4-6 health-related social media posts, which will be posted on our Center's Twitter and Facebook feeds. You will be assigned to post to a feed that is focused on skin health or a feed that is focused on health technologies such as apps and wearables. On Mondays we will remind you to send us your post for the following week as well as the day/time you would like it posted. We will then program your post to appear in our Center's Twitter feed. It will come from our account profile rather than your personal profile. The purpose of the contest is to see which post gets the most engagement. You will receive study compensation for creating each post as well as an opportunity to win the highest engagement gift card weekly. We will give you the names of the Twitter and Facebook feeds to follow so that you can check on your post and others' posts if you wish.

#### Follow-up:

The week after the contest ends (week 5), study staff will email you a link to complete a survey regarding your lifestyle and wellbeing, and your opinion on the contest.

**Time Commitment**: See the table below for the expected time commitment for participating in the study.

| Visit | Time |
|---------------------|--------------|
| | (in minutes) |
| Initial Survey | 5 minutes |
| Telephone Screening | 10 minutes |
| Baseline survey | 15 minutes |
| Webinar | 30 minutes |
| Contest | 1 hour |

| Approx. 10-15 min/week for 4 weeks | |
|------------------------------------|------------|
| Follow-up survey | 30 minutes |
| Total | 2.5 hours |

## What other options are there?

You may choose not to participate in the study.

## What are the risks or inconveniences of the study?

Possible risks related to this research study are: psychological discomfort completing the surveys and personal information could be lost or exposed. To minimize this risk, we will do everything we can to make sure that your information is protected. Confidentiality will be maintained by the use of network secured database and locked file cabinets only accessible to study staff. We also encourage you not to use your name or location in any of the posts that you create.

The Twitter and Facebook feeds that we use are public, which means individuals aside from participants follow it. Your study status as a participant and your identity will not be made known on the Twitter feed. Anything that you comment on, like, or post to the study feed will be extracted and used as study data. This helps us measure the engagement on our feed.

Information you share on Twitter and Facebook is subject to the terms of use and privacy policy, including terms of use for their website and mobile application. You should review these terms and the privacy policy carefully before choosing to download and use the app or use the website. Twitter and Facebook may be able to collect, store and use information about you, such as personal information, location data, shared information, photographs, and more. During the study, if the research team becomes aware of any changes made to privacy policies, we will notify you that this has occurred and will encourage you to review your privacy settings.

For any app or website, we encourage you to choose a password that includes a mix of lowercase letters, uppercase letters, numbers, and symbols, and does not include your username, the app/website name, or other easily-guessable information about you. We also encourage you to not use the same password across different accounts.

Additionally, if you feel discomfort during any part of the study procedures, you may withdraw at any time.

## What are the benefits of the study?

It is hoped that you will receive a benefit of increased awareness of physical and mental wellbeing by participating in this study and taking part in the contest, however we cannot promise a benefit. Benefits to society include providing evidence to support a setting to deliver health and lifestyle messages.

# Will I receive payment for participation? Are there costs to participate?

You will receive \$10 compensation for creating each post (limit of 6 posts). You also have a chance each week to win \$50 if your post receives the most amount of likes, replies and retweets. You will receive extra credit for any posts that get shared. At the end of the study you will

receive \$50 for compensation for completing the follow-up survey. You can also receive \$25 if you refer a friend who ends up joining and completing the study. All compensation will be in the form of emailed Amazon gift cards.

## How will my personal information be protected?

The following procedures will be used to protect the confidentiality of your data. The researchers will keep all study records (including any codes to your data) locked in a secure location on the UConn server. Access to our records will require a UConn login, software login, and personal approval from the program director to access data. At the end of the study, we will remove your name and contact information from the research records and replace with a code. The code will be a three digit number that reflects how many people have contacted the study team to express interest in the study. Data that will be shared with other investigators will be de-identified to help protect your identity. We will remove all identifiable information from the data once the study is complete and extraction data has been analyzed. At this time the link between participant identity and study data will be destroyed. We will keep the de-identified dataset indefinitely. If you end up referring eligible people into the study, or is someone who was referred by another participant, we will protect both parties by not sharing names when discussing any part of the referral process. At the conclusion of this study, the researchers may publish their findings. Information will be presented in summary format and you will not be identified in any publications or presentations.

We will do our best to protect the confidentiality of the information we gather from you but we cannot guarantee 100% confidentiality. Your confidentiality will be maintained to the degree permitted by the technology used. Specifically, no guarantees can be made regarding the interception of data sent via the Internet by any third parties.

You should also know that the UConn Institutional Review Board (IRB) and Research Compliance Services may inspect study records as part of its auditing program, but these reviews will only focus on the researchers and not on your responses or involvement. The IRB is a group of people who review research studies to protect the rights and welfare of research participants.

# Can I stop being in the study and what are my rights?

You do not have to be in this study if you do not want to. If you agree to be in the study, but later change your mind, you may drop out at any time. There are no penalties or consequences of any kind if you decide that you do not want to participate.

# Whom do I contact if I have questions about the study?

Take as long as you like before you make a decision. We will be happy to answer any question you have about this study. If you have further questions about this project or if you have a research-related problem, you may contact the principal investigator, Dr. Sherry Pagoto (sherry.pagoto@uconn.edu, 860-486-2313) or the program director, Jessica Bibeau (jessica.bibeau@uconn.edu, 860-486-8979). If you have any questions concerning your rights as a research subject, you may contact the University of Connecticut Institutional Review Board (IRB) at 860-486-8802.

## **NEXT STEPS**

If you are interested in learning more about this research and participating, proceed to the next page and begin the initial screening survey. In this survey, the only personal contact information we will collect is your email address. If you are eligible to proceed with the study, we will collect

your name and contact information. The questions in this survey will ask questions to determine your eligibility. We will retain this information for our data analysis.

This study is posted on Clinical Trials at: NCT03834974